CLINICAL TRIAL: NCT04182620
Title: Ultrasound-Based Renal Sympathetic Denervation as Adjunctive Upstream Therapy During Atrial Fibrillation Ablation: A Pilot Study
Brief Title: Ultrasound-Based Renal Sympathetic Denervation as Adjunctive Upstream Therapy During Atrial Fibrillation Ablation
Acronym: ULTRA-HFIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 40-5118; IRB 19-02659 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
Keywords: renal denervation; atrial fibrillation; cardiology; electrophysiology
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded until the 6 month visit, at which time they will be un-blinded prior to the follow up CT/MRI. The Clinical Events Committee and Echo Core Lab will remain blinded throughout the trial. In general, the CEC will be blinded to the treatment arms. However, once the nature of the event has been adjudicated, the blind will be broken for that individual patient as necessary to enable the CEC to determine relatedness to the study device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Catheter ablation + renal denervation (Experimental): Catheter ablation + renal denervation
  Interventions: Device: renal denervation; Device: Catheter ablation
- Catheter ablation only (Active Comparator): Catheter ablation
  Interventions: Device: Catheter ablation

INTERVENTIONS:
Device: renal denervation — Renal denervation using the Paradise renal denervation system - a dedicated RDN catheter that delivers a circumferential ring of ablative ultrasound energy
  Arms: Catheter ablation + renal denervation
Device: Catheter ablation — Catheter ablation - one of the most common procedures performed by Cardiac Electrophysiologists for atrial fibrillation

SUMMARY:
The purpose of the ULTRA-HFIB Pilot is to determine the role of adjunctive renal denervation (RDN) in the prevention of Atrial Fibrillation (AF) recurrence in patients scheduled for an AF ablation procedure. Patients will be randomized to either i) AF ablation (Control) or ii) AF ablation + renal sympathetic denervation (Intervention).

DETAILED DESCRIPTION:
The purpose of the ULTRA-HFIB Pilot is to determine the role of adjunctive renal denervation (RDN) in the prevention of AF recurrence in patients scheduled for an AF ablation procedure. Patients will be randomized to either i) AF ablation (Control) or ii) AF ablation + renal sympathetic denervation (Intervention). This is a prospective, controlled, single-blind, randomized trial. The pilot study will be conducted in up to 11 clinical sites in the United States and Europe.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Planned for a first-ever AF ablation procedure (paroxysmal or persistent); (prior to randomization, a technically successful AF ablation procedure, defined as involving pulmonary vein isolation, as well as bidirectional block of any attempted anatomic lesion sets such as cavotricuspid isthmus line, roofline, mitral line and superior vena cava isolation must have been completed)
* History of hypertension and either:

  * Documented history of SBP ≥ 160 or DBP ≥ 100 (Stage III), or
  * Receiving ≥ 1 antihypertensive medication
* Willingness to adhere to study restrictions and comply with all post-procedural follow-up requirements

Exclusion Criteria:

(if any of the following are YES, subject is not eligible)

* Long-standing persistent AF (> 12 months)
* Individual with valvular AF or AF due to a reversible cause
* Prior left atrial catheter or surgical ablation for an atrial arrhythmia (before this index procedure)
* Prior left atrial surgery (such as mitral valve surgery or surgical ASD repair)
* Prior treatment with other devices for hypertension including but not limited to ROX Coupler, Mobius stent and/or the CVRx barostimulator device
* NYHA Class IV Congestive Heart Failure
* Individual has renal artery anatomy that is ineligible for treatment (as determined by intra-procedural renal angiography). This includes:

  * Main renal artery diameter < 3.0 mm or > 8.0 mm
  * Main renal artery length < 20 mm
  * Presence of renal artery stenosis of any origin ≥ 30%
  * Accessory arteries with diameter ≥ 2 mm and < 3.0 mm
  * Calcification in renal arteries at locations where energy is to be delivered
  * Prior renal denervation procedure
  * Presence of abnormal kidney tumors
  * Renal artery aneurysm
  * Pre-existing renal stent or history of renal artery angioplasty
  * Pre-existing aortic stent or history of aortic aneurysm
  * Fibromuscular disease of the renal arteries
  * Iliac/femoral artery stenosis precluding insertion of the Paradise Catheter
* Individual has an estimated glomerular filtration rate (eGFR) of less than 40mL/min/1.73m2
* Inability to undergo AF catheter ablation (e.g., presence of left atrial thrombus, contraindication to all anticoagulation)
* Individual with known allergy to contrast medium not amenable to treatment
* Life expectancy of < 1 year for any medical condition
* Individual has experienced a myocardial infarction, unstable angina, cerebrovascular accident, or heart failure admission within 3 months of screening visit
* Documented history of chronic active inflammatory bowel disorders such as Crohn's disease or ulcerative colitis
* Female participants who are pregnant or nursing
* Individual has known secondary hypertension
* Individual has a single functioning kidney (either congenitally or iatrogenically)
* Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements
* Patients concurrently enrolled in any other investigational drug or device trial that would interfere with the conduction of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Single-procedure freedom from AT/AF/AFL recurrence ≥ 30 seconds | 12 months
  Single-procedure freedom from AT/AF/AFL recurrence ≥ 30 seconds off Class I and III AADs (after the 90-day blanking period), defined by absence of any electrocardiographically documented AT/AF.

SECONDARY OUTCOMES:
Freedom from AT/AF/AFL recurrence | 12 months
  Freedom from AT/AF/AFL recurrence through 12 months (excluding a 90-day blanking period from the initial ablation procedure) irrespective of AADs
Rate of procedural adverse events | 30 days
  Rate of procedural adverse events
The Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) questionnaire | 12 months
  Quality of life instrument (AFEQT) is a 20-item disease-specific scale developed to capture subjective ratings of AF disease and treatment burden. Full range score from 0-100, with higher score indicating higher level of quality of life.
Change in office systolic blood pressure change from baseline to 12 months | 12 months
  Change in office systolic blood pressure change from baseline to 12 months
AF burden at 6 months | 6 months
  AF burden at 6 months
AF burden at 12 months | 12 months
  AF burden at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (13):
- United States (13):
  - University of Arizona - Banner University Medical Center, Phoenix, Arizona
  - Arizona Heart Institute, Phoenix, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Loma Linda University Medical, Loma Linda, California
  - Pacific Heart Institute, Santa Monica, California
  - Hartford Healthcare, Hartford, Connecticut
  - Naples Community Hospital, Naples, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mount Sinai Hospital, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Bellin Memorial Hospital Inc., Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No